CLINICAL TRIAL: NCT06365814
Title: Short- and Long-term Outcomes Following Perioperative ERAS Management in Patients Undergoing Minimally Invasive Radical Gastrectomy After Neoadjuvant Chemotherapy: A Single-center Retrospective Propensity Score Matching Cohort Study
Brief Title: ERAS for Gastric Cancer Patients After NACT
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhouyanbing, Prof., The Affiliated Hospital of Qingdao University
Other Study IDs: ERASforNACT
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS group
  Interventions: Other: enhanced recovery after surgery
- Conventional group
  Interventions: Other: conventional perioperative management

INTERVENTIONS:
Other: enhanced recovery after surgery — ERAS is a comprehensive perioperative interventions, including preoperative patient education, prehabilitation, nutritional support, minimally invasive surgery and other methods, can reduce surgical stress and promote patient recovery
  Groups: ERAS group
Other: conventional perioperative management — conventional perioperative management
  Groups: Conventional group

SUMMARY:
Background: Gastric cancer patients receiving neoadjuvant chemotherapy (NACT) are more vulnerable to perioperative stress. Enhanced recovery after surgery (ERAS) is widely used in surgical patients aiming at reducing stress responses. However, whether this approach is safe and feasible for gastric cancer patients received minimally invasive radical gastrectomy after NACT remained determined. So, the objective of this study is to investigate the effects of ERAS for this special group of gastric cancer patients.

Materials and Methods: The data of gastric cancer patients who underwent minimally invasive radical gastrectomy after NACT were collected in this retrospective cohort study. Patients were divided into an ERAS group and a conventional group based on whether they received perioperative ERAS management. Propensity score matching was conducted to eliminate bias. Pre- and postoperative inflammatory and nutritional marker levels, postoperative complications, recovery indices and 3-year OS and RFS were observed.

DETAILED DESCRIPTION:
Patients From January 2015 to October 2020, the data of 390 gastric cancer patients who underwent laparoscopic or robotic minimally invasive radical gastrectomy after NACT at the Department of Gastrointestinal Surgery, the Affiliated Hospital of Qingdao University, were retrospectively collected and divided into ERAS group and conventional group according to whether they received perioperative ERAS pathway management.

Perioperative management and follow-up Patients in the conventional group received routine perioperative care, while patients in the ERAS group received the ERAS management protocol. Based on clinical practice, we reconsidered the total clauses in the gastric cancer ERAS pathway and determined that preoperative education, prehabilitation, target-oriented liquid management, preoperative oral carbohydrate intake, multimodal analgesia, minimally invasive surgery, physical activity, individual nutritional evaluation and support were the core terms that are suitable for all patients and should be strictly adhered to. Patients follow-up was strictly in accordance with Japanese Gastric Cancer Treatment Guidelines 2021 (6th edition).

NACT and D2 gastrectomy Due to the retrospective design of this study, data from patients who received CapOx, SOX or other 5-fluorouracil-based chemotherapy regimens were collected for analysis. If patients could not complete preoperative chemotherapy as planned due to severe adverse events or if preoperative chemotherapy needed to be prolonged for more than 4 cycles due to unsatisfactory therapeutic efficacy, their data would not be analyzed. If the original regimens were effective before surgery, they were still administered after surgery. If disease progressed after preoperative chemotherapy, subsequent regimens were discussed by a multidisciplinary team. Pre- and postoperative chemotherapy was administered in total of 8 cycles, and this treatment was adjusted according to the patient's disease condition and tolerance.

All patients underwent surgery approximately 4 weeks after the last cycle of preoperative chemotherapy. The extent of gastrectomy was determined according to the tumor location, and the extent of lymph node dissection was strictly in accordance with the D2 standard. The types of digestive tract reconstruction depended on the tumor site, extent of gastric resection, experience and surgeon habits. The choice of laparoscopy or DaVinci-assisted surgery depended on the subjective will of the patients.

Propensity score matching and statistical analysis After excluding patients who did not meet the inclusion criteria, the ERAS group was matched at a ratio of 1:1 with the conventional group including the following covariates: age, PLR, LMR, CAR and prealbumin concentration. SPSS 24.0 was used to perform the match using a 0.2 caliper width.

SPSS 24.0 (IBM, Armonk, NY, USA) was used for the data analysis. The normally distributed measurement data are expressed as mean ± standard deviation (x̅±s); the differences between groups were compared by Student's t test. Measurement data with a nonnormal distribution are presented as medians (interquartile ranges); the Mann-Whitney U test was used for comparisons between two groups. Count data are presented as absolute numbers; comparisons between groups were analyzed using the Chi-square test. The Mann-Whitney U test was used for ranked data. Repeated measures data were analyzed by two-way repeated-measures ANOVA or the generalized estimating equation. Survival curves were plotted using the Kaplan-Meier method, and the differences in survival rate were compared by the log-rank test. Univariate and multivariate analyses of risk factors for RFS and OS were conducted with the Cox proportional hazards regression model. The cutoff values of the continuous variables were determined using the median. The multivariate Cox proportional hazards regression model included variables with p < 0.15 in the univariate analysis. P < 0.05 was considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* gastric adenocarcinoma confirmed by histopathology,
* received 2 to 4 cycles of NACT before surgery,
* minimally invasive (DaVinci or laparoscopy) radical gastrectomy with D2 lymph node dissection

Exclusion Criteria:

* conversion to open surgery due to intraoperative difficulties or uncontrolled complications (for example, intraoperative massive bleeding),
* inability to complete the planned preoperative chemotherapy,
* infeasibility of performing radical gastrectomy during surgery
* ERAS item implementation rate less than 60%

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From January 2015 to October 2020, the data of 390 gastric cancer patients who underwent laparoscopic or robotic minimally invasive radical gastrectomy after NACT at the Department of Gastrointestinal Surgery, the Affiliated Hospital of Qingdao University, were collected and divided into ERAS group and conventional group according to whether they received perioperative ERAS pathway management.
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
postoperative infectious complications | up tp 30 days after surgery
  The primary outcome was the incidence of postoperative infectious complications, which were defined as bacterial infections within 30 d after surgery. The diagnosis of infectious complications was based on fever (≥38°C), elevation of C-reactive protein (CRP), specific clinical symptoms of infection, and positive bacterial culture.

SECONDARY OUTCOMES:
postoperative recovery parameter | up tp 30 days after surgery
  time to first postoperative flatus and bowel movement; time to solid food tolerance; postoperative hospital stay;
blood test result | Postoperative, on postoperative day 1, 3 and 5
  CAR (C-reactive protein-albumin ratio), LMR (lymphocyte-to-monocyte ratio), NLR (neutrophil-to-lymphocyte ratio), PLR (platelet-to-lymphocyte ratio), SII (systemic immune-inflammation index), PNI (prognostic nutrition index), prealbumin and albumin on pre- and postoperative day (POD) 1, 3 and 5 were detected dynamically
3-year overall survival | 3 years
3-years recurrence-free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Surgery, Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided